CLINICAL TRIAL: NCT06559410
Title: A Descriptive Study on Convulsions in Neonates With Congenital Heart Diseases at Assiut University Children Hospital
Brief Title: Convulsions in Neonates With Congenital Heart Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Mohamed Mohamed Abdelhameed, Pediatric resident doctor, Assiut University
Other Study IDs: convulsions in neonates
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Neonatal Convulsion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Electroencephalogram (EEG), CT Brain, Echocardiogram — analyze the etiology, electroencephalographic (EEG) findings, neuroimaging, and neurological sequalae of newborns with congenital heart disease who were presented with seizures

SUMMARY:
analyze the etiology, electroencephalographic (EEG) findings, neuroimaging, and neurological sequalae of newborns with congenital heart disease who were presented with seizures during their neonatal intensive care unit admission.

DETAILED DESCRIPTION:
Neonatal seizures are a commonly encountered neurologic condition in neonates. They are defined as the occurrence of sudden, paroxysmal, abnormal alteration of electrographic activity at any point from birth to the end of the neonatal period. During this period, the neonatal brain is developmentally immature. Thus, neonatal seizures have unique pathophysiology and electrographic findings resulting in clinical manifestations that can be different (and more difficult to identify) when compared to older age groups.

Neonatal seizures are paroxysmal, repetitive and stereotypical events. They are usually clinically subtle, inconspicuous and difficult to recognize from the normal behaviors of the inter-ictal periods or physiological phenomena. There is no recognizable post-ictal state. The most widely used scheme is of five main types of neonatal seizure.

* Subtle seizures (50%)
* Tonic seizures (5%)
* Clonic seizures (25%)
* Myoclonic seizures (20%)
* Non-paroxysmal repetitive behaviors Neonates with congenital heart disease have a high risk of cerebral lesions, seizures, and neurological impairment. By congenital heart disease, we refer to the group of congenital malformations present at birth that include cyanotic as well as non-cyanotic cardiac lesions.

Neonatal seizures are the most common clinical expression of central nervous system dysfunction in newborns and one of the most frequent neurological emergencies during this stage of life. They are usually the first sign of neurological involvement and an indicator of the risk of mortality and/ or neurological sequelae.

ELIGIBILITY:
Inclusion Criteria:

* All neonates up to 28 days of age with congenital heart diseases presented with repeated seizures admitted to Neonatology unit at Assiut university children hospital

Exclusion Criteria:

* Neonates with normal heart or infants more than 28 days of age.

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: neonates with congenital heart diseases
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
analyze the etiology of seizures in newborns with congenital heart disease | baseline
  analyze the etiology of seizures whether it is related to hypoxia, electrolytes disturbances, heart failure or any other casue
analyze the electroencephalographic (EEG) finding and neuroimaging of newborns with congenital heart disease who were presented with seizures | baseline
  neuroimaging including Brain MSCT
state neurological sequalae of newborns with congenital heart disease who were presented with seizures | baseline
  state if there is any neurological sequalae

REFERENCES:
- [Background] Glass HC, Wirrell E. Controversies in neonatal seizure management. J Child Neurol. 2009 May;24(5):591-9. doi: 10.1177/0883073808327832. Epub 2009 Feb 13. PMID 19218527
- [Background] Plouin P, Kaminska A. Neonatal seizures. Handb Clin Neurol. 2013;111:467-76. doi: 10.1016/B978-0-444-52891-9.00051-8. PMID 23622196
- [Background] Abend NS, Wusthoff CJ. Neonatal seizures and status epilepticus. J Clin Neurophysiol. 2012 Oct;29(5):441-8. doi: 10.1097/WNP.0b013e31826bd90d. PMID 23027101
- [Background] Jensen FE. Neonatal seizures: an update on mechanisms and management. Clin Perinatol. 2009 Dec;36(4):881-900, vii. doi: 10.1016/j.clp.2009.08.001. PMID 19944840
- [Background] Proposal for revised classification of epilepsies and epileptic syndromes. Commission on Classification and Terminology of the International League Against Epilepsy. Epilepsia. 1989 Jul-Aug;30(4):389-99. doi: 10.1111/j.1528-1157.1989.tb05316.x. No abstract available. PMID 2502382
- [Background] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Background] Samanek M. Congenital heart malformations: prevalence, severity, survival, and quality of life. Cardiol Young. 2000 May;10(3):179-85. doi: 10.1017/s1047951100009082. No abstract available. PMID 10824896
- [Background] Desnous B, Lenoir M, Doussau A, Marandyuk B, Beaulieu-Genest L, Poirier N, Carmant L, Birca A; CINC multidisciplinary team. Epilepsy and seizures in children with congenital heart disease: A prospective study. Seizure. 2019 Jan;64:50-53. doi: 10.1016/j.seizure.2018.11.011. Epub 2018 Nov 26. PMID 30557820